CLINICAL TRIAL: NCT00591838
Title: A Phase I/II Trial of Stereotactic Body Radiation Therapy (SBRT) Dose Escalation in the Treatment of Patients With Inoperable Stage I/II Non-Small Cell Lung Cancer Arising Within the Zone of the Proximal Bronchial Tree
Brief Title: A Phase I/II Trial of Stereotactic Body Radiation Therapy
Acronym: SBRT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 06-0691 / 201012832
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Inoperable Stage I/II Non-small Cell Lung Cancer
Keywords: SBRT
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Phase I Dose Level A: SBRT 9Gy x 5 fractions (Experimental): -Stereotactic body radiation therapy (SBRT) dose of 9Gy for 5 fractions which is 5 total radiation treatments given over the course of about a week.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Phase I Dose Level B: SBRT 10Gy x 5 fractions (Experimental): -Stereotactic body radiation therapy (SBRT) dose of 10Gy for 5 fractions which is 5 total radiation treatments given over the course of about a week.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Phase I Dose Level C: SBRT 11Gy x 5 fractions (Experimental): -Stereotactic body radiation therapy (SBRT) dose of 11Gy for 5 fractions which is 5 total radiation treatments given over the course of about a week.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Phase I Dose Level D: SBRT 12Gy x 5 fractions (Experimental): -Stereotactic body radiation therapy (SBRT) dose of 12Gy for 5 fractions which is 5 total radiation treatments given over the course of about a week.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Phase II: SBRT 11Gy x 5 fractions (Experimental): -Stereotactic body radiation therapy (SBRT) dose of 11Gy for 5 fractions which is 5 total radiation treatments given over the course of about a week. The phase II dose was determined during the phase I portion of the study.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT)

SUMMARY:
The purpose of this study is to use SBRT in patients with early stage lung cancer and find out what effects (good and bad) SBRT has on their cancer. This research is being done because SBRT has not been used very often in patients with early stage lung cancer or in patients with other serious health problems. In addition, this study also will gather information about patient's health and hospitalization history. This information will be used to find out if there are any factors that can help predict recovery or outcome of patients with lung cancer.

DETAILED DESCRIPTION:
Stage I Non-small Cell Lung Cancer Lung cancer is the most frequent cause of cancer death in both men and women in North America, accounting for approximately 13% of all cancers diagnosed and 28% of all cancer deaths. There will be an estimated 173,770 new lung cancer cases in the United States in the year 2004 with an estimated 160,440 deaths due to lung cancer.1 Seventy-five percent of patients with bronchogenic carcinoma will be diagnosed with non-small cell lung cancer (NSCLC). The number of patients with early or localized disease (currently an estimated 15-20% of NSCLC patients)2 is expected to rise over the next several years due to widespread screening with CT scanning.

The treatment of choice for stage I (T1-T2N0) NSCLC is surgical resection which results in 5-year survival rates of approximately 60 to 70%.3-5 Occasionally, however, there are patients with early-stage NSCLC that are unable to tolerate surgical resection or the postoperative recovery period due to various comorbidities.

While conventionally fractionated radiation therapy has been utilized as nonsurgical therapy for these medically inoperable patients, close observation with no specific cancer therapy has also been advocated in highly selected cases. McGarry, et. al., reviewed outcomes in 75 patients who had received no specific cancer therapy for stage I NSCLC, and the cause of death was progressive cancer in 53% of cases with a median survival time of 14.2 ± 2.4 months.6

Definitive conventionally fractionated RT for early-stage NSCLC is considered reasonable non-surgical therapy but yields poor 5-year survival rates ranging from 10 to 30%.7-11 Several studies have suggested a dose-response relationship reporting a benefit to dose escalation above the standard conventionally fractionated 4,500 to 6,600 cGy. This benefit was evident in both survival and local control in these patients.10-14 Sibley, et. al., reviewed 156 medically inoperable patients with stage I NSCLC treated with primary RT at Duke University between 1980 and 1995. They reported a 5-year, cause-specific survival rate of 32%. There was a trend toward improved survival in those patients achieving local control which approached significance for higher RT doses (p = 0.07).13 At this institution, we have published a series treating 56 patients with medically inoperable NSCLC with a median dose of 70 Gy using conformal radiotherapy techniques.15 Actuarial local control rates were 69% and 63% at two- and three years of follow up, respectively. These data serve as the estimate for statistical power calculations for this trial.

Radiation fields have historically encompassed the primary tumor as well as the regional lymphatics in the ipsilateral hilum and mediastinum. This elective treatment was based on the identified risk of occult lymph node involvement ranging up to 20% in some surgical series.16 In recent years, elimination of elective nodal irradiation, which is potentially poorly tolerated in this population,17 has been validated by several retrospective studies permitting treatment of the primary tumor alone with limited fields.18-21 Slotman, et. al., in a study from the Netherlands, reported the use of limited "postage-stamp" fields to treat early stage lung cancer patients using hypofractionated RT (i.e., 4,800 cGy in 400-cGy fractions). Reported 3-year overall and disease-specific survival rates were 42% and 76%, respectively.20

Most of the aforementioned retrospective studies utilized radiotherapy equipment from the era of 1-D and 2-D treatment planning. Several limitations are evident from these older techniques, including target visualization, selection of beam directions, and computational algorithms describing deposited dose. Recent improvements in software, hardware, and computer processing speed have revolutionized the delivery of radiation doses appropriate for tumor cell killing.

In this new era of three-dimensional treatment planning, more precise delivery methods are available allowing for dose escalation to the target volume without excessive dose being deposited in normal tissues. The RTOG has completed an extensive dose escalation study of conventionally fractionated three-dimensional conformal radiotherapy (3D-CRT) for NSCLC for stages I, II, and III disease as long as all detectable tumor can be encompassed by the radiation therapy fields including both primary tumor and regional lymph nodes.22 No mechanism for minimizing lung and tumor movements was utilized. One hundred and seventy-nine patients were treated with radiation doses escalated to as high as 90.3 Gy. Patients were stratified within each dose level according to the percentage of the total lung volume that received >20 Gy with the treatment plan (V20). For patients receiving radiation alone or radiation following induction chemotherapy, data from RTOG 9311 established that the radiation dose could be safely escalated using 3D-CRT techniques to 83.8 Gy for patients with V20 values of <25% and to 77.4 Gy for patients with V20 values between 25% and 36%, using fraction sizes of 2.15 Gy. Excess mortality was observed at 90.3 Gy with two dose-related deaths. The incidence of grade 3 or higher acute toxicity is less than 10%; however, grade 3 or higher late toxicity was approximately 15%.

Stereotactic Body Radiation Therapy Stereotactic body radiation therapy (SBRT) is the delivery of high precision, biologically potent doses of radiation to tumors of the chest, abdomen, and pelvis. Implementing elements of 3D-CRT with stereotactic targeting, SBRT permits delivery of 3-4 high dose fractions totaling 48-60 Gy with good local control and low toxicity.

A phase I dose escalation trial has been completed at Indiana University for treatment of medically inoperable patients with stage I NSCLC.26, 27 SBRT was administered with large doses per fraction in an extracranial stereotactic body frame, which includes a system for decreasing breathing motion. The starting dose was 8 Gy times 3 (24 Gy total), and fraction dose was escalated by 2 Gy per fraction for each cohort. The target lesion was outlined by a physician and designated as the gross tumor volume (GTV). An additional 0.5 cm in the axial plane and 1.0 cm in the longitudinal plane was added to the GTV to constitute the PTV based on validation measurements for this commercially available system.23, 28, 29 Typically, 7 to 10 non-coplanar beams were used to encompass the PTV. Dose was prescribed to the 80% isodose line. However, higher isodoses occurred within the center of the target mimicking the heterogeneous dose profile common to intracranial stereotactic radiosurgery. The treatment isocenter was identified with 3-D coordinates defined stereotactically and localized on verniers attached to the frame. No skin or bony landmarks were used to set the treatment isocenter; however, orthogonal port films were used on a daily basis for isocenter verification.30 Separate dose escalations were carried out independently for patients with T1 versus T2 small (≤ 5 cm) versus T2 large (5-7 cm) tumors at diagnosis.

According to the Indiana University protocol guidelines, dose-limiting toxicity (DLT) was any grade 3 cardiac or pulmonary toxicity or any grade 4 toxicity attributed to the therapy. Thirty-seven patients were treated using a standard dose escalation protocol with 3 patient cohorts with minimum 1 month between dose levels to assess toxicity. Patients were categorized into separate independent dose escalations according to tumor volume, T1 vs. T2 (≤ 5 cm) vs. T2 (> 5 to ≤ 7 cm). Grade 3 pneumonitis was seen at a dose of 14 x 3 = 42 Gy total in one T2 patient with a 7-cm tumor and transient grade 3 hypoxia was seen at 16 x 3 = 48 Gy total in one patient. Additional patients were treated at each of these levels without further toxicity observed. Twenty-one patients had mild to moderate fibrosis distal to the treated lesion appear on chest x-ray after treatment. Nine of these patients had a decline of an element of their pulmonary function tests (FEV1, FVC, DLCO, or PO2) by 10-20% of predicted which returned back to baseline values with follow-up in all but two. The timing of onset of this toxicity was generally acute to subacute (< 1 month in most cases). The maximum tolerated dose (MTD) was not reached on this trial for patients with T1 tumors and smaller T2 tumors (≤ 5 cm). Dose-limiting pneumonitis or pericarditis occurred in 2/5 patients with larger T2 tumors (>5 to ≤ 7 cm) at a dose of 24 x 3 = 72 Gy defining the MTD for this subgroup at 22 x 3 = 66 Gy. Patients treated at a dose of 22 Gy per fraction times three fractions had follow up of over 24 months without late toxicity for all T-stage tumor categories. Treatment failure within the PTV has been observed in 8 of 26 patients treated at doses of up to 20 x 3 = 60 Gy. However, all but one of these local failures occurred at doses of 16 x 3 = 48 Gy or lower.31

The above data demonstrate that solitary lung lesions including early stage NSCLC are better controlled with SBRT when compared to conventional radiation. In addition, reduced volume treatments are attractive in these patients with medically inoperable stage I NSCLC who may have an increased risk of radiation pneumonitis associated with conventional large volume radiation fields. SBRT permits dose escalation by significantly reducing the high-dose treatment volume.

The RTOG opened in May 2004 a phase II trial of SBRT in the treatment of medically inoperable patients with stage I/II non-small cell lung cancer in an effort to determine if SBRT could achieve acceptable local control as seen in retrospective series.24, 26, 32-38 A secondary objective is to determine if this technique achieves acceptable treatment-related toxicity. In this trial, patients with T1, T2 (≤ 5 cm), or T3 (≤ 5 cm), N0, M0 medically inoperable non-small cell lung cancer are treated with SBRT to a total of 60 Gy in 3 fractions of 20 Gy each over 1.5 to 2 weeks. This protocol excludes patients with T3 tumors involving the central chest and structures of the mediastinum as well as patients with any T-stage tumor within or touching the zone of the proximal bronchial tree. This region is defined as a volume 2 cm in all directions around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus, and right and left lower lobe bronchi).

ELIGIBILITY:
ELIGIBILITY:

Inclusion Criteria

* Histologically confirmed non-small cell cancer by biopsy or cytology. Squamous cell carcinoma, adenocarcinoma, large cell carcinoma, bronchioalveolar carcinoma, or non-small cell carcinoma (not otherwise specified) are allowed.
* Staging studies must identify patient as AJCC Stage I or II based on only 1 of following combinations of TNM staging:

  * T1, N0, M0
  * T2 (<=7cm), N0, M0
  * T3 (<=7cm), N0, M0
* Primary tumor must be arising in one of the following central chest locations:

  * Within or touching the zone of the proximal bronchial tree (a volume 2cm in all directions around the proximal bronchial tree [carina, R & L main bronchi, R & L upper lobe bronchi, intermedius bronchus, R middle lobe bronchus, lingular bronchus, R & L lower lobe bronchi])
  * Adjacent to (within 5 mm) or invading the mediastinal pleura
  * Adjacent to (within 5 mm) or invading the parietal pericardium
* To differentiate T3 lesions involving the mediastinal pleura from T4 lesions involving major vessels or organs, a chest MRI will be obtained. If any uncertainty remains, the patient will have four-dimensional CT scans (4DCT) in an effort to determine the degree of tumor motion. A freely mobile tumor during ventilation will be judged to be T3 disease.
* Patients with hilar or mediastinal lymph nodes <=1cm and no abnormal hilar or mediastinal uptake on PET will be considered N0. Patients with >1cm hilar or mediastinal lymph nodes on CT or abnormal PET (including suspicious but non-diagnostic uptake) may be eligible if directed tissue biopsy of all abnormally identified areas are negative for cancer.
* Primary tumor must be technically resectable by an experienced thoracic cancer clinician, with a reasonable possibility of obtaining a gross total resection with negative margins (potentially curative resection, PCR). However, patients must have underlying physiological medical problems prohibiting PCR (i.e., problems with general anesthesia, the operation, the post-op recovery period, or removal of adjacent functioning lung) or refuse surgery. Deeming a patient medically inoperable based on pulmonary function for surgical resection may include any of the following: baseline FEV1 <40% predicted; post-operative predicted FEV1 <30% predicted; severely reduced diffusion capacity; baseline hypoxemia and/or hypercapnia; exercise oxygen consumption <50% predicted; severe pulmonary hypertension; diabetes with severe end organ damage; severe cerebral, cardiac, or peripheral vascular disease; or severe chronic heart disease. Any one of these problems will qualify a patient for this trial.
* Age >=18.
* Zubrod performance status 0-2.
* Women of childbearing potential must use effective contraception.
* No direct evidence of regional or distant metastases after appropriate staging studies. No synchronous primary or prior malignancy in past 2 years except non-melanoma skin cancer or in situ cancer.
* No previous lung or mediastinal radiation therapy.
* No plans for concomitant antineoplastic therapy (including standard fractionated RT, chemo, biologic, vaccine therapy, or surgery) while on this protocol except at disease progression.
* No active systemic, pulmonary, or pericardial infection.
* No pregnant or lactating women.
* PRESTUDY REQUIREMENTS:

  * History and Physical Examination, Weight, Zubrod performance status (within 4 weeks pre-study entry)
  * Evaluation by thoracic cancer clinician (within 8 weeks pre-study entry)
  * Pregnancy test, if applicable (serum or urine, within 72 hours prior to treatment start.)
  * CT (preferably with contrast unless medically contraindicated; both lungs, mediastinum, liver, adrenals)
  * PET (using FDG with visualization of primary tumor and draining lymph node basins in hilar and mediastinal regions)
  * Brain MRI or head CT with contrast
  * PFTs - include routine spirometry, lung volumes, diffusion capacity
  * Signed informed consent.

Exclusion Criteria:

There is no exclusion criteria associated with this protocol. Please see the above inclusion criteria.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-09-21 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Robinson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levy A, Guckenberger M, Hurkmans C, Nestle U, Belderbos J, De Ruysscher D, Faivre-Finn C, Le Pechoux C. SBRT Dose and Survival in Non-Small Cell Lung Cancer: In Regard to Koshy et al. Int J Radiat Oncol Biol Phys. 2015 Jul 15;92(4):945-6. doi: 10.1016/j.ijrobp.2015.03.032. No abstract available. PMID 26104945
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 09/21/2006 and closed to participant enrollment on 11/01/2017.
Pre-assignment Details: 5 participants in the Phase II portion of study were treated errantly with 10 Gy fractions, rather than 11 Gy fractions, but were included in the analysis as intention-to-treat.
Period: Overall Study
Arm/Group | Phase I Dose Level A: SBRT 9Gy x 5 Fractions | Phase I Dose Level B: SBRT 10Gy x 5 Fractions | Phase I Dose Level C: SBRT 11Gy x 5 Fractions | Phase I Dose Level D: SBRT 12Gy x 5 Fractions | Phase II: SBRT 11Gy x 5 Fractions
Started | 5 | 6 | 6 | 6 | 51
Completed | 5 | 6 | 6 | 5 | 51
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level A: SBRT 9Gy x 5 Fractions | Phase I Dose Level B: SBRT 10Gy x 5 Fractions | Phase I Dose Level C: SBRT 11Gy x 5 Fractions | Phase I Dose Level D: SBRT 12Gy x 5 Fractions | Phase II: SBRT 11Gy x 5 Fractions | Total
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 51 | 74
Age, Continuous [Median (Full Range); unit: years] | 71 [62 to 82] | 79.5 [64 to 87] | 78 [62 to 87] | 73.5 [62 to 85] | 73 [52 to 89] | 74.5 [52 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 4 | 23 | 29
  Male | 4 | 6 | 5 | 2 | 28 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 0 | 2 | 5 | 6 | 50 | 63
  Unknown or Not Reported | 4 | 4 | 1 | 0 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 4 | 1 | 3 | 0 | 8 | 16
  White | 1 | 4 | 0 | 5 | 39 | 49
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 3 | 0 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 6 | 6 | 51 | 74

OUTCOME MEASURES:

1. Primary Outcome: Phase I Portion Only: Determine the Maximum Tolerated Dose of SBRT
Description: The phase 1 portion had a "5+3" strategy with four escalating dose levels, only one of which was open for accrual at any time. Five patients were accrued to each dose level, and once closed, the next dose level could not be opened until the preceding dose was deemed acceptable. With a minimum of 90 days from the start of RT, if there were no acute grade 3 or 4 non-hematologic toxicities in the five patients, the current dose was deemed acceptable. If one such toxicity was observed, an additional 3 patients were recruited and followed for a minimum of 90 days. If 2 or more such toxicities were observed, the current dose was determined as dose limiting, and the previous dose level was used for the phase 2 portion.
Time Frame: Completion of phase I enrollment (Phase I enrollment took 4 years)
Population: Phase I participants were the only participants evaluable for this outcome measure
Measure: Number; unit: Gy x 5 fractions
Groups:
- Phase I: Stereotactic Body Radiation (SBRT): SBRT
  Dose Level A 9Gy x 5 fractions
  Dose Level B 10 Gy x 5 fractions
  Dose Level C 11 Gy x 5 fractions
  Dose Level D 12 Gy x 5 fractions
Arm/Group | Phase I: Stereotactic Body Radiation (SBRT)
Number analyzed (Participants) | 22
Gy x 5 fractions | 11

2. Primary Outcome: Phase I Portion Only: Number of Participants With Acute Treatment Related Grade 3-5 Toxicity
Description: * CTCAE version 3.0 will be used to grade toxicity
  * Acute toxicity are adverse events that occur from start of treatment through 90 days
Time Frame: Up to 90 days
Population: -Phase I participants were the only evaluable participants for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level A: SBRT 9Gy x 5 Fractions | Phase I Dose Level B: SBRT 10Gy x 5 Fractions | Phase I Dose Level C: SBRT 11Gy x 5 Fractions | Phase I Dose Level D: SBRT 12Gy x 5 Fractions
Number analyzed (Participants) | 5 | 6 | 6 | 6
Participants
  Lymphopenia | 0 | 1 | 0 | 0
  Neutrophils/granulocytes (ANC/AGC) | 0 | 1 | 0 | 0
  Glucose, serum-high (hyperglycemia) | 0 | 1 | 0 | 0
  Sodium, serum-low (hyponatremia) | 0 | 1 | 0 | 0
  Arthritis (non-septic) | 0 | 1 | 0 | 0
  Cataract | 1 | 0 | 0 | 0
  Dyspnea (shortness of breath) | 0 | 1 | 0 | 1
  Flu-like syndrome | 0 | 0 | 0 | 1

3. Primary Outcome: Phase I Portion Only: Number of Participants With Late Treatment Related Grade 3-5 Toxicity
Description: * CTCAE version 3.0 will be used to grade toxicity
  * Late toxicity are adverse events that occur from Day 91 through 2 years
Time Frame: 91 days to 2 years
Population: -Phase I participants were the only participants evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level A: SBRT 9Gy x 5 Fractions | Phase I Dose Level B: SBRT 10Gy x 5 Fractions | Phase I Dose Level C: SBRT 11Gy x 5 Fractions | Phase I Dose Level D: SBRT 12Gy x 5 Fractions
Number analyzed (Participants) | 5 | 6 | 6 | 6
Participants
  Atrial fibrillation | 0 | 0 | 1 | 0
  Prolonged QTc interval | 0 | 0 | 1 | 0
  Pneumonia | 0 | 2 | 2 | 2
  Generalized weakness | 0 | 0 | 0 | 0
  Chest/thorax NOS pain | 0 | 0 | 1 | 0
  Hypoxia | 0 | 0 | 1 | 0
  Cough | 0 | 0 | 1 | 0
  Dyspnea | 1 | 3 | 4 | 2
  Pneumonitis/pulmonary infiltrates | 0 | 0 | 1 | 1

4. Primary Outcome: Phase II Portion Only: Local Control Rate
Description: Local control rate is defined as the absence of isolated failure (progression) within the primary tumor and involved lobe
Time Frame: 2 years
Population: Phase I participants were not evaluable for this outcome measure. 1 patient in Phase II did not come back for follow-up. The remaining 50 participants were analyzed for the outcome measure but only those who were not lost to follow-up or deceased at 2 years were included in the outcome measure results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: SBRT 11Gy x 5 Fractions
Number analyzed (Participants) | 50
percentage of participants | 85 [62 to 95]

5. Secondary Outcome: Phase II Only: Regional Nodal Recurrence Rate
Description: Regional nodal recurrence is defined as absence of isolated failure (progression) within hilar/mediastinal/supraclavicular lymph nodes.
Time Frame: 2 years
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Phase II: SBRT 11Gy x 5 Fractions
Number analyzed (Participants) | 50
percentage of participants | 0

6. Secondary Outcome: Phase II Only: Disseminated Recurrence Rate
Description: Disseminated recurrence is defined as the absence of failure (progression) outside ipsilateral lung and hilar/mediastinal/supraclavicular lymph nodes.
Time Frame: 2 years
Population: Phase I participants were not evaluable for this outcome measure. 1 patient in Phase II did not come back for follow-up and was excluded from analysis. The remaining 50 participants were analyzed for the outcome measure but only those who were not lost to follow-up or deceased at 2 years were included in the outcome measure results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: SBRT 11Gy x 5 Fractions
Number analyzed (Participants) | 50
percentage of participants | 27 [15 to 45]

7. Secondary Outcome: Phase II Only: Disease-free Survival Rate
Description: Disease-free survival rate is defined as patients without any disease failure (progression), second primary, or death from any cause.
Time Frame: 2 years
Population: Phase I participants were excluded from this outcome measure. 1 patient in Phase II did not come back for follow-up and was excluded from analysis. The remaining 50 participants were analyzed for the outcome measure but only those who were not lost to follow-up or deceased at 2 years were included in the outcome measure results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: SBRT 11Gy x 5 Fractions
Number analyzed (Participants) | 50
percentage of participants | 28 [16 to 42]

8. Secondary Outcome: Phase II Only: Overall Survival Rate
Description: Overall survival is defined as patients alive
Time Frame: 2 years
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: SBRT 11Gy x 5 Fractions
Number analyzed (Participants) | 50
percentage of participants | 43 [28 to 57]

ADVERSE EVENTS:
Time Frame: Acute adverse events from protocol radiation therapy was collected from start of treatment until 90 days. Late adverse events from protocol radiation therapy was collected from day 91 until completion of follow-up. Mean follow-up for Dose Level A=22.9 months (full range 6-47), Dose Level B=25.3 months (full range 2-42), Dose Level C=17.3 months (full range 13-22), Dose Level D 6.6 months (full range 1-11), Phase II=17 months (full range 2-57).
Description: Grade 2 or above acute and late adverse events from protocol radiation therapy were collected. For purposes of this protocol, serious adverse events related to stereotactic radiation therapy include those listed as Grade 3-5 within the CTCAE document. All-cause mortality was followed from start of treatment until completion of follow-up or death, whichever came first.
Arm/Group | Phase I Dose Level A: SBRT 9Gy x 5 Fractions | Phase I Dose Level B: SBRT 10Gy x 5 Fractions | Phase I Dose Level C: SBRT 11Gy x 5 Fractions | Phase I Dose Level D: SBRT 12Gy x 5 Fractions | Phase II: SBRT 11Gy x 5 Fractions
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/6 | 2/6 | 3/6 | 35/51
Serious Adverse Events (participants affected / at risk) | 1/5 | 3/6 | 4/6 | 4/6 | 23/51
Other Adverse Events (participants affected / at risk) | 3/5 | 3/6 | 4/6 | 3/6 | 32/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level A: SBRT 9Gy x 5 Fractions (N=5) | Phase I Dose Level B: SBRT 10Gy x 5 Fractions (N=6) | Phase I Dose Level C: SBRT 11Gy x 5 Fractions (N=6) | Phase I Dose Level D: SBRT 12Gy x 5 Fractions (N=6) | Phase II: SBRT 11Gy x 5 Fractions (N=51)
Acute - Lymphopenia (Investigations) | 0 | 1 | 0 | 0 | 1
Acute - Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 | 1 | 0 | 0 | 0
Acute - Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Acute - Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Acute - Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Acute - Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Acute - Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Acute - Flu-like syndrome (General disorders) | 0 | 0 | 0 | 0 | 0
Late - Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Late - Prolonged QTc interval (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Late - Pneumonia (Infections and infestations) | 0 | 2 | 2 | 2 | 11
Late - Generalized weakness (General disorders) | 0 | 1 | 0 | 1 | 2
Late - Chest/thorax NOS pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Late - Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 6
Late - Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 6
Late - Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 2 | 13
Late - Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 3
Acute - Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Acute - Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Acute - Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Acute - Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acute - Infection, Other (Urinary tract infection) (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acute - AST, SGOT (Investigations) | 0 | 0 | 0 | 0 | 1
Acute - Creatinine (Investigations) | 0 | 0 | 0 | 0 | 1
Acute - Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Acute - Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Acute - Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Acute - Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Acute - Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Acute - Prolonged intubation thru pulmonary resection (>24 hours thru surgery) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Late - Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Late - Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Late - Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Late - Port site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Late - Bronchospasm/wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Late - Obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Late - Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Late - Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level A: SBRT 9Gy x 5 Fractions (N=5) | Phase I Dose Level B: SBRT 10Gy x 5 Fractions (N=6) | Phase I Dose Level C: SBRT 11Gy x 5 Fractions (N=6) | Phase I Dose Level D: SBRT 12Gy x 5 Fractions (N=6) | Phase II: SBRT 11Gy x 5 Fractions (N=51)
Acute - Hemoglobin (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 4
Acute - Lymphopenia (Investigations) | 1 | 0 | 0 | 0 | 2
Acute - Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1
Acute - Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Acute - Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2
Acute - Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Late - Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0 | 3
Late - Generalized weakness (General disorders) | 0 | 0 | 0 | 1 | 1
Late - Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3
Late - Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 4
Late - Chest/thorax NOS pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 5
Late - Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 6
Late - Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 10
Late - Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 7
Late - Obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Late - Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 6
Acute - Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Acute - Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Acute - Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Acute - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Acute - Infection, Other (shingles, sepsis) (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acute - Albumin, serum-low (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Acute - Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Acute - Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
Acute - Pain - chest wall (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
Acute - Pain - shoulder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Acute - Acelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Acute - Carbon monoxide diffusion capacity (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acute - Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Acute - Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Acute - FEV(1) (Investigations) | 0 | 0 | 0 | 0 | 1
Acute - Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Late - Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Late - Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Late - Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Late - Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Late - Bronchospasm/wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Late - Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT00591838/Prot_SAP_000.pdf